CLINICAL TRIAL: NCT00961753
Title: Safety and Efficacy of an Optimized Ibuprofen Dosing Regimen Versus Standard Dosing for Pharmacologic Closure of Patent Ductus Arteriosus
Brief Title: Safety/Efficacy Study of Optimizing Ibuprofen Dosing to Achieve Higher PDA Closure Rates
Acronym: OIDS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA drug recall on July 30, 2010
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, James Hocker, M.D., OSF Healthcare System
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ibuprofendosingstudy
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; Ibuprofen; Preterm; Neonate
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimized Ibuprofen (Experimental)
  Interventions: Drug: optimized ibuprofen
- Standard Ibuprofen (Active Comparator)
  Interventions: Drug: Standard Ibuprofen

INTERVENTIONS:
Drug: optimized ibuprofen — day of life 0-3 - 10, 5, 5 mg/kg/dose at 24 hour intervals day of life 4-6 - 14, 7, 7 mg/kg/dose at 24 hour intervals day of life 7-29 - 20, 10, 10 mg/kg/dose at 24 hour intervals
  Other Names: neoprofen
  Arms: Optimized Ibuprofen
Drug: Standard Ibuprofen — day of life 0-29 - 10,5, 5 mg/kg/dose at 24 hour intervals
  Other Names: neoprofen
  Arms: Standard Ibuprofen

SUMMARY:
The purpose of this study is to determine if increasing the ibuprofen dose will increase the likelihood of closing the patent ductus arteriosus in premature babies.

DETAILED DESCRIPTION:
Failure to close the PDA in premature neonates in a timely fashion can lead to pulmonary over-circulation and systemic under-circulation. The PDA often fails to close using currently approved Ibuprofen dosing regimens, and surgical closure becomes necessary. Ibuprofen clearance in premature neonates is significantly correlated with postnatal age, increasing rapidly over time. Hirt et al. published and optimized dosing scheme for preterm neonates based on pharmacokinetic and pharmacodynamic data. We aim to use this dosing regimen in the clinical setting to determine if increased rates of pharmacologic PDA closure can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* All neonates (0-29 days old) less than or equal to 33 post-menstrual age at time of PDA diagnosis requiring nasal CPAP or mechanical ventilation
* Echo confirmed PDA with a transductal diameter of 1.5 mm or greater and demonstrating a left-to-right shunt
* Signed informed consent

Exclusion Criteria:

* Presence of: ductal-dependent congenital heart disease, pulmonary hypertension,
* Active bleeding (including Grade 3 or 4 IVH)
* Platelet count < 100,000
* Coagulopathy
* Suspected NEC
* Suspected perforation
* Creatinine > 1.5
* Hyperbilirubinemia requiring exchange transfusion
* Hypotension requiring pressor support
* Life-threatening congenital malformation

Ages: 1 Day to 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
PDA Closure | 1-42 days of age

SECONDARY OUTCOMES:
renal function | 1-30 days of age

CONTACTS AND LOCATIONS:
Overall Officials: James R Hocker, MD, Principal Investigator — OSF Healthcare System
Locations (1):
- Children's Hospital of Illinois at OSF Saint Francis Medical Center, Peoria, Illinois, United States